CLINICAL TRIAL: NCT03439670
Title: A Phase IIb Randomized, Double-blind, Parallel Group, Placebo- and Active-controlled Study With Double-Blind Extension to Assess the Efficacy and Safety of Vamorolone in Ambulant Boys With Duchenne Muscular Dystrophy (DMD)
Brief Title: A Study to Assess the Efficacy and Safety of Vamorolone in Boys With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Collaborators: European Union (Other); Cooperative International Neuromuscular Research Group (Network); Newcastle University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBP15-004
Record Dates: First submitted 2018-01-09; First posted 2018-02-20 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Vamorolone
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — VBP15 compound; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Treatment Group 1 (Experimental): Patients enrolled in Treatment Group 1 (experimental group) will receive vamorolone 2.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Group 2 (Experimental): Patients enrolled in Treatment Group 2 (experimental group) will receive vamorolone at 6.0 mg/kg/day for the duration of the study.
  Interventions: Drug: Vamorolone
- Treatment Group 3 (Active Comparator): Patients enrolled in Treatment Group 3 (active comparator group) will receive prednisone 0.75 mg/kg/day for 24 weeks followed by 20 weeks of treatment with 2.0 mg/kg/day vamorolone.
  Interventions: Drug: Prednisone; Drug: Vamorolone
- Treatment Group 4 (Active Comparator): Patients enrolled in Treatment Group 4 (active comparator group) will receive prednisone 0.75 mg/kg/day for 24 weeks followed by 20 weeks treatment with 6.0 mg/kg/day vamorolone.
  Interventions: Drug: Prednisone; Drug: Vamorolone
- Treatment Group 5 (Placebo Comparator): Patients enrolled in Treatment Group 5 (placebo comparator group) will receive placebo daily for 24 weeks followed by 20 weeks treatment with 2.0 mg/kg/day vamorolone.
  Interventions: Other: Placebo; Drug: Vamorolone
- Treatment Group 6 (Placebo Comparator): Patients enrolled in Treatment Group 6 (placebo comparator group) will receive placebo daily for 24 weeks followed by 20 weeks treatment with 6.0 mg/kg/day vamorolone.
  Interventions: Other: Placebo; Drug: Vamorolone

INTERVENTIONS:
Drug: Vamorolone — Oral administration of 2.0 mg/kg/day for the duration of the study.
  Other Names: VBP15
  Arms: Treatment Group 1
Drug: Prednisone — Oral administration of 0.75 mg/kg/day for 24 weeks.
  Arms: Treatment Group 3
Other: Placebo — Oral administration of placebo daily for 24 weeks.
  Arms: Treatment Group 5
Drug: Vamorolone — Oral administration of 6.0 mg/kg/day for the duration of the study.
  Other Names: VBP15
  Arms: Treatment Group 2
Drug: Prednisone — Oral administration of 0.75 mg/kg/day for 24 weeks.
  Arms: Treatment Group 4
Other: Placebo — Oral administration of placebo daily for 24 weeks.
  Arms: Treatment Group 6
Drug: Vamorolone — Oral administration of 2.0 mg/kg/day for 20 weeks.
  Other Names: VBP15
  Arms: Treatment Group 3; Treatment Group 5
Drug: Vamorolone — Oral administration of 6.0 mg/kg/day for 20 weeks.
  Other Names: VBP15
  Arms: Treatment Group 4; Treatment Group 6

SUMMARY:
Brief Summary: This Phase IIb study is a randomized, double-blind, parallel group, placebo and active-controlled study to evaluate the efficacy, safety, PD, and population PK of vamorolone administered orally at daily doses of 2.0 mg/kg and 6.0 mg/kg versus prednisone 0.75 mg/kg/day and placebo over a Treatment Period of 24 weeks, and to evaluate persistence of effect over a Treatment Period of 48 weeks in ambulant boys ages 4 to <7 years with DMD.

DETAILED DESCRIPTION:
This Phase IIb study is a randomized, double-blind, parallel group, placebo and active-controlled study to evaluate the efficacy, safety, PD, and population PK of vamorolone administered orally at daily doses of 2.0 mg/kg and 6.0 mg/kg versus prednisone 0.75 mg/kg/day and placebo over a Treatment Period of 24 weeks, and to evaluate persistence of effect over a Treatment Period of 48 weeks in ambulant boys ages 4 to <7 years with DMD.

The study is comprised of a 5-week Pretreatment Screening Period, a 1-day Pretreatment Baseline Period, a 24-week Treatment Period #1 (Weeks 1-24), a 4-week Transition Period (Weeks 25-28), a 20-week Treatment Period #2 (Weeks 28 + 1 day to 48), and a 4-week Dose-tapering Period (Weeks 49-52).

Subjects will be randomized to one of six treatment groups in a 2:2:1:1:1:1 ratio, where the two prednisone groups in Treatment Period #1 (Groups 3 and 4) will be combined and the two placebo groups in Treatment Period #1 (Groups 5 and 6) will be combined, effectively resulting in a 1:1:1:1 randomization (vamorolone 2.0 mg/kg/day : vamorolone 6.0 mg/kg/day : prednisone 0.75 mg/kg/day : placebo) for Treatment Period #1.

Subjects will be stratified based on age at study entry (<6 vs. ≥ 6 years). During the 4-week Transition Period between Treatment Period #1 and Treatment Period #2, all subjects will continue on the same oral suspension (vamorolone 2.0 mg/kg or 6.0 mg/kg, or matching placebo) they received during Treatment Period #1 and all subjects will have their tablet dose tapered to zero. Thus, subjects randomized to receive vamorolone during Treatment Period #1 (Groups 1 and 2) will continue to receive vamorolone at the same dose, while subjects randomized to receive prednisone will have their dose tapered to zero, and subjects randomized to placebo will continue to receive placebo.

The prednisone group will be used as an active control comparison for safety and efficacy endpoints as requested by the European Medicines Agency (EMA). The placebo group will be used as comparator for efficacy endpoints (superiority model) as requested by the EMA and Food and Drug Administration (FDA) protocol advisory board. Although glucocorticoids are part of the care recommendations for DMD, their adverse effect profile has limited their use. The age at which glucocorticoids should be started in DMD boys is uncertain, ranging from 4 to 7 years, based on a balance between benefits and side effects. In view of the age inclusion criteria and duration of the placebo-controlled study period (6 months), the use of a placebo group has been considered acceptable as in clinical practice it will not cause a real delay in prescription of an accepted treatment for this condition. Any exposure of placebo longer than 6 months was considered unethical.

At the end of the Treatment Period #2, subjects may be given access to vamorolone through an additional study or general access program, or given the option to transition to standard of care treatment for DMD (may include glucocorticoids). Subjects completing VBP15-004 and enrolling directly into an additional vamorolone study or general access program to receive vamorolone will not need to taper their vamorolone dose prior to enrollment. All other subjects will begin a 4-week double-blind Dose-tapering Period during which the dose of study medication will be progressively reduced and discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's parent(s) or legal guardian(s) has (have) provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, where applicable, prior to any study-related procedures; participants will be asked to give written or verbal assent according to local requirements
2. Subject has a centrally confirmed (by TRiNDS central genetic counselor[s]) diagnosis of DMD as defined as:

   * Dystrophin immunofluorescence and/or immunoblot showing complete dystrophin deficiency, and clinical picture consistent with typical DMD, OR
   * Identifiable mutation within the DMD gene (deletion/duplication of one or more exons), where reading frame can be predicted as 'out-of-frame,' and clinical picture consistent with typical DMD, OR
   * Complete dystrophin gene sequencing showing an alteration (point mutation, duplication, other) that is expected to preclude production of the dystrophin protein (i.e., nonsense mutation, deletion/duplication leading to a downstream stop codon), with a clinical picture consistent with typical DMD;
3. Subject is ≥ 4 years and <7 years of age at time of enrollment in the study;
4. Subject weighs >13.0 kg and ≤ 39.9 kg at the Screening Visit;
5. Subject is able to walk independently without assistive devices;
6. Subject is able to complete the Time to Stand Test (TTSTAND) without assistance in <10 seconds, as assessed at the Screening Visit;
7. Clinical laboratory test results are within the normal range at the Screening Visit, or if abnormal, are not clinically significant, in the opinion of the Investigator. [Notes: Serum gamma glutamyl transferase (GGT), creatinine, and total bilirubin all must be ≤ upper limit of the normal range at the Screening Visit. An abnormal vitamin D level that is considered clinically significant will not exclude a subject from randomization];
8. Subject has evidence of chicken pox immunity as determined by:

   * Presence of IgG antibodies to varicella, as documented by a positive test result from the local laboratory from blood collected during the Screening Period, OR
   * Documentation, provided at the Screening Visit, that the subject has had 2 doses of varicella vaccine, with or without serologic evidence of immunity; the second of the 2 immunizations must have been given at least 14 days prior to randomization.
9. Subject is able to swallow tablets, as confirmed by successful test swallowing of placebo tablets during the Screening Period; and
10. Subject and parent(s)/guardian(s) are willing and able to comply with scheduled visits, study drug administration plan, and study procedures.

Exclusion Criteria:

1. Subject has current or history of major renal or hepatic impairment, diabetes mellitus or immunosuppression;
2. Subject has current or history of chronic systemic fungal or viral infections;
3. Subject has had an acute illness within 4 weeks prior to the first dose of study medication;
4. Subject has used mineralocorticoid receptor agents, such as spironolactone, eplerenone, canrenone (canrenoate potassium), prorenone (prorenoate potassium), mexrenone (mexrenoate potassium) within 4 weeks prior to the first dose of study medication;
5. Subject has a history of primary hyperaldosteronism;
6. Subject has evidence of symptomatic cardiomyopathy [Note: Asymptomatic cardiac abnormality on investigation would not be exclusionary];
7. Subject is currently being treated or has received previous treatment with oral glucocorticoids or other immunosuppressive agents [Notes: Past transient use of oral glucocorticoids or other oral immunosuppressive agents for no longer than 1 month cumulative, with last use at least 3 months prior to first dose of study medication, will be considered for eligibility on a case-by-case basis, unless discontinued for intolerance. Inhaled and/or topical glucocorticoids are permitted if last use is at least 4 weeks prior to first dose of study medication or if administered at stable dose beginning at least 4 weeks prior to first dose of study medication and anticipated to be used at the stable dose regimen for the duration of the study];
8. Subject has an allergy or hypersensitivity to the study medication or to any of its constituents;
9. Subject has used idebenone within 4 weeks prior to the first dose of study medication;
10. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the Investigator;
11. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow-up will be correctly completed or impair the assessment of study results, in the opinion of the Investigator;
12. Subject is taking (or has taken within 4 weeks prior to the first dose of study medication) herbal remedies and supplements which can impact muscle strength and function (e.g., Co-enzyme Q10, creatine, etc);
13. Subject is taking (or has taken within 3 months prior to the first dose of study medication) any medication indicated for DMD, including Exondys51 and Translarna;
14. Subject has been administered a live attenuated vaccine within 14 days prior to the first dose of study medication;
15. Subject is currently taking any other investigational drug or has taken any other investigational drug within 3 months prior to the first dose of study medication;
16. Subject has a sibling who is currently enrolled in any vamorolone study or Expanded Access Program, or who intends to enroll in any vamorolone study or Expanded Access Program during the subject's participation in the VBP15-004 study; or
17. Subject has previously been enrolled in the study. Note: Any parameter/test may be repeated at the Investigator's discretion during Screening to determine reproducibility. In addition, subjects may be rescreened if ineligible due to a transient condition which would prevent the subject from participating, such as an upper respiratory tract infection or injury, or if ineligible due to negative anti-varicella IgG antibody test result.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michela Guglieri, M.D., Study Chair — John Walton Muscular Dystrophy Research Centre; Paula Clemens, M.D., Study Chair — University of Pittsburgh
Locations (33):
- United States (10):
  - University of California Davis, Davis, California
  - University of California Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Nemours Children's Hospital, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Gillette Children's Speciality Health Care, Saint Paul, Minnesota
  - Duke Children's Hospital, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of Virginia of Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Royal Children's Hospital, Melbourne
  - Sydney Children's Hospital, Westmead
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Hospitals Leuven, Leuven
- Canada (4):
  - Alberta's Children Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Czechia (2):
  - University Hospital Brno, Brno
  - Charles University, Prague
- Agia Sofia Children's Hospital, Athens, Greece
- Schneider Children's Medical Center, Petah Tikvah, Israel
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud University, Nijmegen
- Spain (2):
  - Sant Joan de Deu Hospital - Barcelona, Spain, Barcelona
  - Hospital Universitario y Politécnico La Fe, Valencia
- Queen Silvia Children's Hospital, Gothenburg, Sweden
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Hospital for Children, Glasgow
  - Leeds Teaching Hospital Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Background] Mah JK, Korngut L, Dykeman J, Day L, Pringsheim T, Jette N. A systematic review and meta-analysis on the epidemiology of Duchenne and Becker muscular dystrophy. Neuromuscul Disord. 2014 Jun;24(6):482-91. doi: 10.1016/j.nmd.2014.03.008. Epub 2014 Mar 22. PMID 24780148
- [Background] Hoffman EP, Brown RH Jr, Kunkel LM. Dystrophin: the protein product of the Duchenne muscular dystrophy locus. Cell. 1987 Dec 24;51(6):919-28. doi: 10.1016/0092-8674(87)90579-4. PMID 3319190
- [Background] Evans NP, Misyak SA, Robertson JL, Bassaganya-Riera J, Grange RW. Immune-mediated mechanisms potentially regulate the disease time-course of duchenne muscular dystrophy and provide targets for therapeutic intervention. PM R. 2009 Aug;1(8):755-68. doi: 10.1016/j.pmrj.2009.04.010. PMID 19695529
- [Background] Kumar A, Boriek AM. Mechanical stress activates the nuclear factor-kappaB pathway in skeletal muscle fibers: a possible role in Duchenne muscular dystrophy. FASEB J. 2003 Mar;17(3):386-96. doi: 10.1096/fj.02-0542com. PMID 12631578
- [Background] Acharyya S, Villalta SA, Bakkar N, Bupha-Intr T, Janssen PM, Carathers M, Li ZW, Beg AA, Ghosh S, Sahenk Z, Weinstein M, Gardner KL, Rafael-Fortney JA, Karin M, Tidball JG, Baldwin AS, Guttridge DC. Interplay of IKK/NF-kappaB signaling in macrophages and myofibers promotes muscle degeneration in Duchenne muscular dystrophy. J Clin Invest. 2007 Apr;117(4):889-901. doi: 10.1172/JCI30556. Epub 2007 Mar 22. PMID 17380205
- [Background] Dogra C, Changotra H, Wergedal JE, Kumar A. Regulation of phosphatidylinositol 3-kinase (PI3K)/Akt and nuclear factor-kappa B signaling pathways in dystrophin-deficient skeletal muscle in response to mechanical stretch. J Cell Physiol. 2006 Sep;208(3):575-85. doi: 10.1002/jcp.20696. PMID 16741926
- [Background] Pahl HL. Activators and target genes of Rel/NF-kappaB transcription factors. Oncogene. 1999 Nov 22;18(49):6853-66. doi: 10.1038/sj.onc.1203239. PMID 10602461
- [Background] Spencer MJ, Montecino-Rodriguez E, Dorshkind K, Tidball JG. Helper (CD4(+)) and cytotoxic (CD8(+)) T cells promote the pathology of dystrophin-deficient muscle. Clin Immunol. 2001 Feb;98(2):235-43. doi: 10.1006/clim.2000.4966. PMID 11161980
- [Background] Spencer MJ, Tidball JG. Do immune cells promote the pathology of dystrophin-deficient myopathies? Neuromuscul Disord. 2001 Sep;11(6-7):556-64. doi: 10.1016/s0960-8966(01)00198-5. PMID 11525885
- [Background] Malik V, Rodino-Klapac LR, Mendell JR. Emerging drugs for Duchenne muscular dystrophy. Expert Opin Emerg Drugs. 2012 Jun;17(2):261-77. doi: 10.1517/14728214.2012.691965. PMID 22632414
- [Background] Reeves EKM, Hoffman EP, Nagaraju K, Damsker JM, McCall JM. VBP15: preclinical characterization of a novel anti-inflammatory delta 9,11 steroid. Bioorg Med Chem. 2013 Apr 15;21(8):2241-2249. doi: 10.1016/j.bmc.2013.02.009. Epub 2013 Feb 18. PMID 23498916
- [Background] Bushby K, Finkel R, Birnkrant DJ, Case LE, Clemens PR, Cripe L, Kaul A, Kinnett K, McDonald C, Pandya S, Poysky J, Shapiro F, Tomezsko J, Constantin C; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and pharmacological and psychosocial management. Lancet Neurol. 2010 Jan;9(1):77-93. doi: 10.1016/S1474-4422(09)70271-6. Epub 2009 Nov 27. PMID 19945913
- [Background] Pane M, Mazzone ES, Sivo S, Sormani MP, Messina S, D'Amico A, Carlesi A, Vita G, Fanelli L, Berardinelli A, Torrente Y, Lanzillotta V, Viggiano E, D Ambrosio P, Cavallaro F, Frosini S, Barp A, Bonfiglio S, Scalise R, De Sanctis R, Rolle E, Graziano A, Magri F, Palermo C, Rossi F, Donati MA, Sacchini M, Arnoldi MT, Baranello G, Mongini T, Pini A, Battini R, Pegoraro E, Previtali S, Bruno C, Politano L, Comi GP, Bertini E, Mercuri E. Long term natural history data in ambulant boys with Duchenne muscular dystrophy: 36-month changes. PLoS One. 2014 Oct 1;9(10):e108205. doi: 10.1371/journal.pone.0108205. eCollection 2014. PMID 25271887
- [Background] Manzur AY, Kuntzer T, Pike M, Swan A. Glucocorticoid corticosteroids for Duchenne muscular dystrophy. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD003725. doi: 10.1002/14651858.CD003725.pub3. PMID 18254031
- [Background] Heier CR, Damsker JM, Yu Q, Dillingham BC, Huynh T, Van der Meulen JH, Sali A, Miller BK, Phadke A, Scheffer L, Quinn J, Tatem K, Jordan S, Dadgar S, Rodriguez OC, Albanese C, Calhoun M, Gordish-Dressman H, Jaiswal JK, Connor EM, McCall JM, Hoffman EP, Reeves EK, Nagaraju K. VBP15, a novel anti-inflammatory and membrane-stabilizer, improves muscular dystrophy without side effects. EMBO Mol Med. 2013 Oct;5(10):1569-85. doi: 10.1002/emmm.201302621. Epub 2013 Sep 9. PMID 24014378
- [Background] Damsker JM, Dillingham BC, Rose MC, Balsley MA, Heier CR, Watson AM, Stemmy EJ, Jurjus RA, Huynh T, Tatem K, Uaesoontrachoon K, Berry DM, Benton AS, Freishtat RJ, Hoffman EP, McCall JM, Gordish-Dressman H, Constant SL, Reeves EK, Nagaraju K. VBP15, a glucocorticoid analogue, is effective at reducing allergic lung inflammation in mice. PLoS One. 2013 May 7;8(5):e63871. doi: 10.1371/journal.pone.0063871. Print 2013. PMID 23667681
- [Background] Dillingham BC, Knoblach SM, Many GM, Harmon BT, Mullen AM, Heier CR, Bello L, McCall JM, Hoffman EP, Connor EM, Nagaraju K, Reeves EKM, Damsker JM. VBP15, a novel anti-inflammatory, is effective at reducing the severity of murine experimental autoimmune encephalomyelitis. Cell Mol Neurobiol. 2015 Apr;35(3):377-387. doi: 10.1007/s10571-014-0133-y. Epub 2014 Nov 13. PMID 25392236
- [Background] Dadgar S, Wang Z, Johnston H, Kesari A, Nagaraju K, Chen YW, Hill DA, Partridge TA, Giri M, Freishtat RJ, Nazarian J, Xuan J, Wang Y, Hoffman EP. Asynchronous remodeling is a driver of failed regeneration in Duchenne muscular dystrophy. J Cell Biol. 2014 Oct 13;207(1):139-58. doi: 10.1083/jcb.201402079. PMID 25313409
- [Background] Raman SV, Hor KN, Mazur W, Halnon NJ, Kissel JT, He X, Tran T, Smart S, McCarthy B, Taylor MD, Jefferies JL, Rafael-Fortney JA, Lowe J, Roble SL, Cripe LH. Eplerenone for early cardiomyopathy in Duchenne muscular dystrophy: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2015 Feb;14(2):153-61. doi: 10.1016/S1474-4422(14)70318-7. Epub 2014 Dec 30. PMID 25554404
- [Background] Avioli LV. Glucocorticoid effects on statural growth. Br J Rheumatol. 1993 May;32 Suppl 2:27-30. doi: 10.1093/rheumatology/32.suppl_2.27. PMID 8495277
- [Background] Wolthers OD, Pedersen S. Short term linear growth in asthmatic children during treatment with prednisolone. BMJ. 1990 Jul 21;301(6744):145-8. doi: 10.1136/bmj.301.6744.145. PMID 2202451
- [Background] Bircan Z, Soran M, Yildirim I, Dogan M, Sahin A, Bilici A, Danaci M. The effect of alternate-day low dose prednisolone on bone age in children with steroid dependent nephrotic syndrome. Int Urol Nephrol. 1997;29(3):357-61. doi: 10.1007/BF02550936. PMID 9285311
- [Background] Manolagas SC, Weinstein RS. New developments in the pathogenesis and treatment of steroid-induced osteoporosis. J Bone Miner Res. 1999 Jul;14(7):1061-6. doi: 10.1359/jbmr.1999.14.7.1061. No abstract available. PMID 10404005
- [Background] Sali A, Guerron AD, Gordish-Dressman H, Spurney CF, Iantorno M, Hoffman EP, Nagaraju K. Glucocorticoid-treated mice are an inappropriate positive control for long-term preclinical studies in the mdx mouse. PLoS One. 2012;7(4):e34204. doi: 10.1371/journal.pone.0034204. Epub 2012 Apr 3. PMID 22509280
- [Background] Kauh E, Mixson L, Malice MP, Mesens S, Ramael S, Burke J, Reynders T, Van Dyck K, Beals C, Rosenberg E, Ruddy M. Prednisone affects inflammation, glucose tolerance, and bone turnover within hours of treatment in healthy individuals. Eur J Endocrinol. 2012 Mar;166(3):459-67. doi: 10.1530/EJE-11-0751. Epub 2011 Dec 17. PMID 22180452
- [Background] Wehling-Henricks M, Oltmann M, Rinaldi C, Myung KH, Tidball JG. Loss of positive allosteric interactions between neuronal nitric oxide synthase and phosphofructokinase contributes to defects in glycolysis and increased fatigability in muscular dystrophy. Hum Mol Genet. 2009 Sep 15;18(18):3439-51. doi: 10.1093/hmg/ddp288. Epub 2009 Jun 19. PMID 19542095
- [Background] Younes M, Neffati F, Touzi M, Hassen-Zrour S, Fendri Y, Bejia I, Ben Amor A, Bergaoui N, Najjar MF. Systemic effects of epidural and intra-articular glucocorticoid injections in diabetic and non-diabetic patients. Joint Bone Spine. 2007 Oct;74(5):472-6. doi: 10.1016/j.jbspin.2006.10.009. Epub 2007 Jul 6. PMID 17919959
- [Background] Moon HJ, Choi KH, Lee SI, Lee OJ, Shin JW, Kim TW. Changes in blood glucose and cortisol levels after epidural or shoulder intra-articular glucocorticoid injections in diabetic or nondiabetic patients. Am J Phys Med Rehabil. 2014 May;93(5):372-8. doi: 10.1097/PHM.0000000000000001. PMID 24508924
- [Background] Investigator's Brochure, Version 4, Vamorolone (17α,21-dihydroxy-16α-methyl-pregna-1,4,9(11)-triene-3,20-dione) 4% Oral Suspension, ReveraGen BioPharma, Inc., January 10, 2017.
- [Background] Fleishaker DL, Mukherjee A, Whaley FS, Daniel S, Zeiher BG. Safety and pharmacodynamic dose response of short-term prednisone in healthy adult subjects: a dose ranging, randomized, placebo-controlled, crossover study. BMC Musculoskelet Disord. 2016 Jul 16;17:293. doi: 10.1186/s12891-016-1135-3. PMID 27424036
- [Background] Hathout Y, Conklin LS, Seol H, Gordish-Dressman H, Brown KJ, Morgenroth LP, Nagaraju K, Heier CR, Damsker JM, van den Anker JN, Henricson E, Clemens PR, Mah JK, McDonald C, Hoffman EP. Serum pharmacodynamic biomarkers for chronic corticosteroid treatment of children. Sci Rep. 2016 Aug 17;6:31727. doi: 10.1038/srep31727. PMID 27530235
- [Background] Agwu JC, Spoudeas H, Hindmarsh PC, Pringle PJ, Brook CG. Tests of adrenal insufficiency. Arch Dis Child. 1999 Apr;80(4):330-3. doi: 10.1136/adc.80.4.330. PMID 10086937
- [Background] van Staa TP, Leufkens HG, Abenhaim L, Zhang B, Cooper C. Oral corticosteroids and fracture risk: relationship to daily and cumulative doses. Rheumatology (Oxford). 2000 Dec;39(12):1383-9. doi: 10.1093/rheumatology/39.12.1383. PMID 11136882
- [Background] McDonald C, Camino E, Escandon R, Finkel RS, Fischer R, Flanigan K, Furlong P, Juhasz R, Martin AS, Villa C, Sweeney HL. Draft Guidance for Industry Duchenne Muscular Dystrophy, Becker Muscular Dystrophy, and Related Dystrophinopathies - Developing Potential Treatments for the Entire Spectrum of Disease. J Neuromuscul Dis. 2024;11(2):499-523. doi: 10.3233/JND-230219. PMID 38363616
- [Background] Brooke MH, Griggs RC, Mendell JR, Fenichel GM, Shumate JB, Pellegrino RJ. Clinical trial in Duchenne dystrophy. I. The design of the protocol. Muscle Nerve. 1981 May-Jun;4(3):186-97. doi: 10.1002/mus.880040304. No abstract available. PMID 7017401
- [Background] Mazzone ES, Messina S, Vasco G, Main M, Eagle M, D'Amico A, Doglio L, Politano L, Cavallaro F, Frosini S, Bello L, Magri F, Corlatti A, Zucchini E, Brancalion B, Rossi F, Ferretti M, Motta MG, Cecio MR, Berardinelli A, Alfieri P, Mongini T, Pini A, Astrea G, Battini R, Comi G, Pegoraro E, Morandi L, Pane M, Angelini C, Bruno C, Villanova M, Vita G, Donati MA, Bertini E, Mercuri E. Reliability of the North Star Ambulatory Assessment in a multicentric setting. Neuromuscul Disord. 2009 Jul;19(7):458-61. doi: 10.1016/j.nmd.2009.06.368. Epub 2009 Jun 23. PMID 19553120
- [Background] McDonald CM, Henricson EK, Han JJ, Abresch RT, Nicorici A, Elfring GL, Atkinson L, Reha A, Hirawat S, Miller LL. The 6-minute walk test as a new outcome measure in Duchenne muscular dystrophy. Muscle Nerve. 2010 Apr;41(4):500-10. doi: 10.1002/mus.21544. PMID 19941337
- [Background] Bello L, Kesari A, Gordish-Dressman H, Cnaan A, Morgenroth LP, Punetha J, Duong T, Henricson EK, Pegoraro E, McDonald CM, Hoffman EP; Cooperative International Neuromuscular Research Group Investigators. Genetic modifiers of ambulation in the Cooperative International Neuromuscular Research Group Duchenne Natural History Study. Ann Neurol. 2015 Apr;77(4):684-96. doi: 10.1002/ana.24370. Epub 2015 Mar 13. PMID 25641372
- [Background] Spurney C, Shimizu R, Morgenroth LP, Kolski H, Gordish-Dressman H, Clemens PR; CINRG Investigators. Cooperative International Neuromuscular Research Group Duchenne Natural History Study demonstrates insufficient diagnosis and treatment of cardiomyopathy in Duchenne muscular dystrophy. Muscle Nerve. 2014 Aug;50(2):250-6. doi: 10.1002/mus.24163. Epub 2014 May 14. PMID 24395289
- [Background] McDonald CM, Henricson EK, Abresch RT, Han JJ, Escolar DM, Florence JM, Duong T, Arrieta A, Clemens PR, Hoffman EP, Cnaan A; Cinrg Investigators. The cooperative international neuromuscular research group Duchenne natural history study--a longitudinal investigation in the era of glucocorticoid therapy: design of protocol and the methods used. Muscle Nerve. 2013 Jul;48(1):32-54. doi: 10.1002/mus.23807. Epub 2013 May 16. PMID 23677550
- [Background] Henricson EK, Abresch RT, Cnaan A, Hu F, Duong T, Arrieta A, Han J, Escolar DM, Florence JM, Clemens PR, Hoffman EP, McDonald CM; CINRG Investigators. The cooperative international neuromuscular research group Duchenne natural history study: glucocorticoid treatment preserves clinically meaningful functional milestones and reduces rate of disease progression as measured by manual muscle testing and other commonly used clinical trial outcome measures. Muscle Nerve. 2013 Jul;48(1):55-67. doi: 10.1002/mus.23808. Epub 2013 May 6. PMID 23649481
- [Background] Escolar DM, Hache LP, Clemens PR, Cnaan A, McDonald CM, Viswanathan V, Kornberg AJ, Bertorini TE, Nevo Y, Lotze T, Pestronk A, Ryan MM, Monasterio E, Day JW, Zimmerman A, Arrieta A, Henricson E, Mayhew J, Florence J, Hu F, Connolly AM. Randomized, blinded trial of weekend vs daily prednisone in Duchenne muscular dystrophy. Neurology. 2011 Aug 2;77(5):444-52. doi: 10.1212/WNL.0b013e318227b164. Epub 2011 Jul 13. PMID 21753160
- [Result] Guglieri M, Clemens PR, Perlman SJ, Smith EC, Horrocks I, Finkel RS, Mah JK, Deconinck N, Goemans N, Haberlova J, Straub V, Mengle-Gaw LJ, Schwartz BD, Harper AD, Shieh PB, De Waele L, Castro D, Yang ML, Ryan MM, McDonald CM, Tulinius M, Webster R, McMillan HJ, Kuntz NL, Rao VK, Baranello G, Spinty S, Childs AM, Sbrocchi AM, Selby KA, Monduy M, Nevo Y, Vilchez-Padilla JJ, Nascimento-Osorio A, Niks EH, de Groot IJM, Katsalouli M, James MK, van den Anker J, Damsker JM, Ahmet A, Ward LM, Jaros M, Shale P, Dang UJ, Hoffman EP. Efficacy and Safety of Vamorolone vs Placebo and Prednisone Among Boys With Duchenne Muscular Dystrophy: A Randomized Clinical Trial. JAMA Neurol. 2022 Oct 1;79(10):1005-1014. doi: 10.1001/jamaneurol.2022.2480. PMID 36036925
- [Derived] de Vera A, Clemens PR, Dang UJ, Dutreix C, Gresko E, Guglieri M, Hagerty L, Hasham S, Damsker J, Hathout Y, Linden A, Berglund A, Tobin R, Wahbi K, Hoffman EP. Mineralocorticoid receptor antagonism of vamorolone: Evidence from LIONHEART and VISION-DMD clinical trials. Steroids. 2025 Nov;223:109689. doi: 10.1016/j.steroids.2025.109689. Epub 2025 Sep 14. PMID 40957504
- [Derived] Dang UJ, Damsker JM, Guglieri M, Clemens PR, Perlman SJ, Smith EC, Horrocks I, Finkel RS, Mah JK, Deconinck N, Goemans NM, Haberlova J, Straub V, Mengle-Gaw L, Schwartz BD, Harper A, Shieh PB, De Waele L, Castro D, Yang ML, Ryan MM, McDonald CM, Tulinius M, Webster RI, Mcmillan HJ, Kuntz N, Rao VK, Baranello G, Spinty S, Childs AM, Sbrocchi AM, Selby KA, Monduy M, Nevo Y, Vilchez JJ, Nascimento-Osorio A, Niks EH, De Groot IJM, Katsalouli M, Van Den Anker JN, Ward LM, Leinonen M, D'Alessandro AL, Hoffman EP. Efficacy and Safety of Vamorolone Over 48 Weeks in Boys With Duchenne Muscular Dystrophy: A Randomized Controlled Trial. Neurology. 2024 Mar 12;102(5):e208112. doi: 10.1212/WNL.0000000000208112. Epub 2024 Feb 9. PMID 38335499

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group 1: Patients enrolled in Treatment Group 1 (experimental group) will receive vamorolone 2.0 mg/kg/day for 24 weeks followed by vamorolone 2.0mg/kg/day for 20 weeks.
- Treatment Group 2: Patients enrolled in Treatment Group 2 (experimental group) will receive vamorolone 6.0 mg/kg/day for 24 weeks followed by vamorolone 6.0mg/kg/day for 20 weeks.
- Treatment Group 3: Patients enrolled in Treatment Group 3 (active comparator group) will receive prednisone 0.75 mg/kg/day for 24 weeks followed by vamorolone 2.0mg/kg/day for 20 weeks.
- Treatment Group 4: Patients enrolled in Treatment Group 4 (active comparator group) will receive prednisone 0.75 mg/kg/day for 24 weeks followed by vamorolone 6.0mg/kg/day for 20 weeks.
- Treatment Group 5: Patients enrolled in Treatment Group 5 will receive placebo for 24 weeks followed by vamorolone 2mg/kg/day for 20 weeks.
- Treatment Group 6: Patients enrolled in Treatment Group 6 will receive placebo for 24 weeks followed by vamorolone 6mg/kg/day for 20 weeks.
Period: Overall Study
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
Started | 30 | 30 | 15 | 16 | 15 | 15
Completed | 28 | 26 | 15 | 15 | 14 | 14
Not Completed | 2 | 4 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population refers to the baseline visit per protocol while the Participant Flow refers to all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Total
Number analyzed (Participants) | 28 | 28 | 15 | 15 | 14 | 14 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 28 | 15 | 15 | 14 | 14 | 114
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 28 | 28 | 15 | 15 | 14 | 14 | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 4 | 3 | 2 | 1 | 1 | 1 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 23 | 23 | 12 | 12 | 11 | 13 | 94
  More than one race | 0 | 1 | 1 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
TTSTAND (seconds) [Mean (Standard Deviation); unit: Seconds] | 6.01 (2.406) | 5.97 (1.991) | 5.36 (1.948) | 4.53 (0.808) | 5.51 (1.578) | 5.58 (2.288) | 5.560 (1.9498)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measured by Time to Stand Test (TTSTAND) Velocity in Rises/Second Change From Baseline
Description: Vamorolone at 6.0mg/kg/day vs. placebo group in change from baseline to the Week 24 assessment
Time Frame: 24 weeks
Population: Per the protocol, the primary clinical efficacy endpoint was "comparison of the vamorolone 6.0 mg/kg/day dose level group versus the placebo group in change from baseline to the Week 24 assessment."
Measure: Mean (Standard Deviation); unit: Rises/Seconds
Groups:
- Treatment Group 1: Patients enrolled in Treatment Group 1 (placebo comparator group) will receive placebo for 24 weeks.
- Treatment Group 2: Patients enrolled in Treatment Group 2 (experimental group) will receive vamorolone 6.0 mg/kg/day for 24 weeks
Arm/Group | Treatment Group 1 | Treatment Group 2
Number analyzed (Participants) | 28 | 27
Rises/Seconds | -.007 (0.0628) | 0.054 (0.0666)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/15 | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/28 | 2/28 | 0/15 | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 26/28 | 26/28 | 15/15 | 13/15 | 12/14 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (N=28) | Treatment Group 2 (N=28) | Treatment Group 3 (N=15) | Treatment Group 4 (N=15) | Treatment Group 5 (N=14) | Treatment Group 6 (N=14)
Gastroenteritis viral/viral gasteroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group 1 (N=28) | Treatment Group 2 (N=28) | Treatment Group 3 (N=15) | Treatment Group 4 (N=15) | Treatment Group 5 (N=14) | Treatment Group 6 (N=14)
Abdominal Pain (Gastrointestinal disorders) | 3 | 3 | 2 | 1 | 2 | 0
Abdominal Pain upper (Gastrointestinal disorders) | 1 | 3 | 3 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 3 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 6 | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 7 | 3 | 3 | 1 | 3 | 3
Gasteroenteritis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3 | 2 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 10 | 4 | 2 | 3 | 3 | 2
Rhinitis (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 4 | 2 | 3 | 0 | 1
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1
Protein Urine Present (Investigations) | 1 | 0 | 1 | 3 | 0 | 0
Weight increased (Investigations) | 1 | 3 | 1 | 1 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1 | 1 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 4 | 2 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 1 | 0 | 3
Psychomotor hyperactivity (Nervous system disorders) | 2 | 0 | 1 | 2 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 2 | 1 | 2 | 0 | 1 | 1
Aggression (Psychiatric disorders) | 2 | 1 | 0 | 2 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 3 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 2 | 4 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2 | 0 | 0
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 2 | 1 | 2
Mouth Ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulance (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enterobiasis (Infections and infestations) | 1 | 2 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Ear Infection (Infections and infestations) | 1 | 1 | 0 | 1 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 1
Tonsilitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral/viral gasteroenteritis (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0
Moluscum contagiosum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Otitis media bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Respiratory track infection viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Steptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 4 | 9 | 4 | 4 | 1 | 1
Growth hormone deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ligament strain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1
Athralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Costrochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertebral wedging (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Agitation (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 1 | 0
Anger (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Dysphemia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Enuresis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Oppositional defiant disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Trichotillomania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epistaxis (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0
Night sweats (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash macropapular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Viral rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cortisol decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 1
Bacterial test postive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lipase decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 2 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 1 | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT03439670/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03439670/SAP_003.pdf